CLINICAL TRIAL: NCT01585077
Title: Comparison of the Susceptibility of Naive and Pre-immune Volunteers to Infectious Challenge With Viable Plasmodium Vivax Sporozoites.
Brief Title: Exposure of Naive and Pre-immune Subjects to P. Vivax Challenge
Acronym: ChallengeIII
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Socrates Herrera Valencia (Other)
Responsible Party: Sponsor-Investigator, Socrates Herrera Valencia, Director, Malaria Vaccine and Drug Development Center
Organization: Malaria Vaccine and Drug Development Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CIV - 08 - 102010
Record Dates: First submitted 2012-04-23; First posted 2012-04-25 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Malaria
Keywords: Plasmodium vivax; Malaria; Challenge; Anopheles albimanus
MeSH Terms: conditions — Malaria; Malaria, Vivax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naive volunteers (Experimental): Volunteers without previous exposure to malaria, and negative antibody titers (<1:20) against native protein of P. vivax.
  Interventions: Biological: P. vivax infected mosquito bites
- Pre-immune volunteers (Experimental): Volunteers with previous exposure to malaria, and positive antibody titers against native protein of P. vivax
  Interventions: Biological: P. vivax infected mosquito bites

INTERVENTIONS:
Biological: P. vivax infected mosquito bites — All volunteers will receive one dose of 2-4 P. vivax infected mosquito bites. All the mosquitoes will correspond to the same mosquito batch to make sure that all volunteers receive the same P. vivax strain.

SUMMARY:
This study is a randomized clinical trial designed to compare the susceptibility of naive and pre-immune volunteers to infectious challenge with viable Plasmodium vivax sporozoites. The term preimmune hereafter denoted only previous experience with infection by this parasite and not a definite state of immunity to malaria infection. The study hypothesis is that pre-immune volunteers present a delayed onset of malaria clinical and parasitological manifestations when compared to naive individuals. The development of this study will establish a protocol for evaluating the effectiveness of vaccine candidates against P. vivax in subsequent Phases IIa and IIb clinical trials.

DETAILED DESCRIPTION:
This study is a prospective controlled, blinded clinical trial, designed to establish the differences on infectivity of an infectious challenge with P. vivax sporozoites between human volunteers with and without history of malaria.

Study subjects

This study will require the involvement of two types of volunteers:

- Parasite donors: 5-15 P. vivax-infected patients who will serve as parasites donors for experimental infection of mosquitoes, who will be enrolled in the endemic area.

- Volunteers for infectious challenge Two other groups of volunteers will be exposed to mosquitoes infected with P. vivax sporozoites. A group of 7 people without previous exposure to malaria (naive) and another 12 people with a history of previous malaria infection (pre-immune).

Methodology

* Recruitment of infected patients Parasite donors will be recruited among P. vivax infected patients attending a diagnostic center in the endemic area.
* Infection of mosquitoes Blood from donors will be used to feed three days old mosquitoes by artificial membrane feeding technique. At day 7 a sample of mosquitoes will be examined to determine the degree of infection by dissection of the mosquito gut. On day 14, a small amount of mosquitoes with a good degree of infectivity will be used to infect challenged volunteers.
* Recruitment of pre-immune and naive volunteers Volunteers for the challenge will be recruited both in the city of Cali, non-endemic region, and in Buenaventura, a malaria endemic region, through various activities such as conferences, meetings and other means approved by the IRB like posters and flyers.

Infection of volunteers

The "feeding cage" will be placed on the forearm of a volunteer for 10 minutes, allowing that the feeding window, wich will be covered by a mesh surface be placed against the volunteer's skin.

Follow Up

Volunteers will be educated about the signs and symptoms of malaria and they will have a daily telephone contact during the first 6 days.

Between days 7 and 23 the volunteers will be asked to go to the Clinical Trials Unit daily in order to establish the presence or absence of disease through thick blood smear and samples will be collected for retrospective real time PCR P. vivax.

From day 23 until day 31, volunteers will receive physical and laboratory evaluation every other day and will have daily telephone contact.

Once the patients present signs and symptoms of the disease curative treatment will be immediately provided, and 15 ml of blood will be drawn, which will be used for immune response assessment.

If the volunteers do not develop the disease during the follow-up period, on day 31 they will be given antimalarial treatment.

Treatment

Volunteers will be treated with antimalarial drugs approved by the Colombian Ministry of Social Protection: chloroquine (three (3) doses: 600 mg initially, followed by 450mg at 24, and 48 hours), associated with primaquine (30mg/día) for 14 days. All the volunteers will be asked to return two weeks after starting treatment for a thick blood smear test to ensure cure of malaria.

ELIGIBILITY:
Inclusion Criteria:

1. Step 1:

   * Age 15 to 60 years.
   * Hemoglobin levels > 9g/dL.
   * Presence of Current P. vivax infection.
   * Absence of other Plasmodium species determined by thick blood smear and PCR.
   * Blood parasite count of 0.1% or more.
   * Absence of other acute or chronic diseases.
   * Being able to sign an informed consent form.
2. Step 2:

   * Healthy 18 to 45 years old man or non-pregnant women.
   * To have the capacity to sign an informed consent in a free and voluntary way.
   * To have an acceptable understanding of the clinical trial through the approval of a questionnaire regarding the information given in the consent process.
   * Obligatory use of adequate contraceptive method from beginning of recruitment and screening time up to three months after last immunization.
   * Do not have chronic or acute diseases. These conditions will be determined by clinical history, physical exam and laboratory tests.
   * To accept not traveling to malaria endemic areas during the clinical trial should
   * To have telephone at home or mobile phone that permit permanent contact for follow up
   * Being willing to participated during both steps of the clinical trial.

Exclusion Criteria:

1. Step 1:

   * history of blood transfusion in the last six months.
   * Pregnancy in women.
   * Have received antimalarial treatment before the diagnosis.
2. Step 2:

   * Pregnant or nursing women.
   * History of moderate or severe insect, or food allergies.
   * G-6PD deficiency or any Hb genetic defect.
   * Symptoms, signs or data from laboratory test that suggests any systemic disorder like renal, hepatic, cardiovascular, pulmonary, psychiatric disorders or other illnesses that could interfere with results of clinical trial or could compromise the health of the volunteer.
   * To have antibodies against hepatitis C, VIH, or hepatitis B superficial antigen and/or hepatitis B core antibodies.
   * To have any abnormality in the parameters assessed by blood laboratory tests
   * Presence or history of an auto-immune disease.
   * History of surgical removal of the spleen (splenectomy).
   * Use of medical treatment known to alter the immune system before 3 months to recruitment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pre-patent period onset | Two months after the challenge
  begining at day 7 after mosquito bites exposure, both groups of volunteers will be evaluated with dayly Thick blood smear to compare the malaria onset between the pre-immune and naive groups.

SECONDARY OUTCOMES:
Immune response | Two months after the malaria challenge
  Malaria signs and symptoms will be assessed to stablish severity and frequency of appearence in both groups: Pre-immune and naive.
  Blood sample will be taken at the end of the study to determine the differences in celular and humoral immune responses in both study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sócrates Herrera, MD, Principal Investigator — Malaria Vaccine and Drug Development Center
Locations (1):
- Malaria Vaccine and Drug development Center (MVDC), Cali, Valle del Cauca Department, Colombia

REFERENCES:
- [Background] Herrera S, Solarte Y, Jordan-Villegas A, Echavarria JF, Rocha L, Palacios R, Ramirez O, Velez JD, Epstein JE, Richie TL, Arevalo-Herrera M. Consistent safety and infectivity in sporozoite challenge model of Plasmodium vivax in malaria-naive human volunteers. Am J Trop Med Hyg. 2011 Feb;84(2 Suppl):4-11. doi: 10.4269/ajtmh.2011.09-0498. PMID 21292872
- [Background] Herrera S, Fernandez O, Manzano MR, Murrain B, Vergara J, Blanco P, Palacios R, Velez JD, Epstein JE, Chen-Mok M, Reed ZH, Arevalo-Herrera M. Successful sporozoite challenge model in human volunteers with Plasmodium vivax strain derived from human donors. Am J Trop Med Hyg. 2009 Nov;81(5):740-6. doi: 10.4269/ajtmh.2009.09-0194. PMID 19861603
- [Derived] Arevalo-Herrera M, Forero-Pena DA, Rubiano K, Gomez-Hincapie J, Martinez NL, Lopez-Perez M, Castellanos A, Cespedes N, Palacios R, Onate JM, Herrera S. Plasmodium vivax sporozoite challenge in malaria-naive and semi-immune Colombian volunteers. PLoS One. 2014 Jun 25;9(6):e99754. doi: 10.1371/journal.pone.0099754. eCollection 2014. PMID 24963662
- See also: Malaria Vaccine and Drug Development Center web page — http://www.inmuno.org